CLINICAL TRIAL: NCT02991781
Title: Multidisciplinary Tools for Improving the Efficacy of Public Prevention Measures Against Smoking
Brief Title: Combined Bio- and Neuro- Feedback vs. Varenicline Use for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: AAI Scientific Cultural Services Ltd (AAISCS) (Other); NATIONAL ASSOCIATION OF GENERAL PRACTITIONERS IN BULGARIA (Unknown)
Responsible Party: Principal Investigator, Panos Bamidis, Dr. Panagiotis Bamidis, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SEP-210254111
Record Dates: First submitted 2015-05-05; First posted 2016-12-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Smoking | interventions — Biofeedback, Psychology; Neurofeedback; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- COPD Patients (Experimental): C.O.P.D. patients: Presence of a post-bronchodilator forced expiratory volume at one second (FEV1) / forced vital capacity (FVC) < 0.70 with symptoms as dyspnea, chronic cough, chronic sputum production
  Biofeedback and Neurofeedback Training
  Varenicline use for smoking cessation
  Passive Control
  Interventions: Other: Biofeedback and Neurofeedback Training; Drug: Varenicline use for smoking cessation; Other: Passive Control
- Asthma Patients (Experimental): Asthma patients: Presence of 2 or more of symptoms of airflow obstruction (cough, wheezing, dyspnea). Airflow obstruction at least partially reversible demonstrated by spirometry with FEV1 increased by >12% following b2 agonist inhalation) or evidence of bronchial hyperresponsiveness by metacholine provocation test (demonstrated by provocative concentration causing a 20% fall (PC20) <8 mg or mannitol provocation test (with FEV1 decrease of 15%)
  Biofeedback and Neurofeedback Training
  Varenicline use for smoking cessation
  Passive Control
  Interventions: Other: Biofeedback and Neurofeedback Training; Drug: Varenicline use for smoking cessation; Other: Passive Control
- Smokers (Experimental): Smokers will consist of a group of patients that are under the age of 35, unemployed and healthy according to a standard clinical evaluation.
  Biofeedback and Neurofeedback Training
  Varenicline use for smoking cessation
  Sham Neurofeedback
  Passive Control
  Interventions: Other: Biofeedback and Neurofeedback Training; Drug: Varenicline use for smoking cessation; Other: Sham Neurofeedback; Other: Passive Control

INTERVENTIONS:
Other: Biofeedback and Neurofeedback Training — The protocol will consist of 5 sessions of skin temperature biofeedback and 20 sessions of a neurofeedback training protocol that will consist of Alpha-Theta ratio up-training. The aim of the training is to reach a crossover state, were initially Alpha activity will increase and then in a deeper state, the Theta activity will take over. This state is associated with a reverie and disidentification with problems, stress or traumatic experiences. Therefore, the subjects will learn how to increase their Theta/Alpha ratio.
  Other Names: Neurofeedback
Drug: Varenicline use for smoking cessation — The protocol will consist 1 mg varenicline use twice daily following a 1-week titration for 3 months.
  Other Names: Varenicline
Other: Sham Neurofeedback — Subjects will receive equal sessions of sham neurofeedback, and thus serve as a control group for the analysis and design of the study.
  Other Names: Active Control
  Arms: Smokers
Other: Passive Control — Subjects will not receive any intervention, but they will be measured via a clinical and psychometric evaluation with a time-difference of 3 months. This is equal to the intervention time. Hence, the subjects in this intervention type will serve as a control group for the analysis and design of the study.

SUMMARY:
This study will develop and experimentally test the efficiency of a neurofeedback training protocol vs. varenicline use for smoking cessation.

DETAILED DESCRIPTION:
This study will develop and experimentally test the efficiency of a neurofeedback(NF) training protocol for smoking cessation. As non-pharmacological, non-invasive and painless brainwave technique, NF contributes to teach individuals how they can take the control of their mind through operant conditioning. NF regulates brain function in natural way. Studies have reported an 80% rate of reducing or eliminating the need for traditional medication14. Therefore, other nicotine substitutes (such as varenicline) which may carry their own toxicity risk factor may become redundant. The protocol will include 5 bio- and 25 Neuro-feedback sessions, lasting approximately 36 months.

The electrophysiological evaluation of the efficacy of the intervention will include EEG resting state and a multifeature Mismatch Negativity (MMN) evoked response measurements before and after the participation of human volunteers. These data will be analyzed in terms of cortical activation patterns and cortical connectivity. Questionnaires will be used to collect behavioral and psychometric data regarding smoking related behaviors. Additionally, a clinical evaluation including spirometry, exhaled carbon monoxide, total antioxidant capacity, vitamine E, and cotinine will be conducted. The data will be collected prior, during, after the completion of the study and after a one-year follow up.

The Neurofeedback intervention will be compared to a different group of participants that will follow an intervention based on varenicline use for approximately 3 months. The electrophysiological evaluation of the efficacy of the intervention will include EEG resting state and a sleep polysomnography measurement. Questionnaires and clinical evaluation include the same measurements as the neurofeedback intervention but only in 3 time points: prior, during, after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being continuous tobacco smokers (>10 cigarettes per day) for at least 6 months
* Being unemployed for at least 3 months
* Being diagnosed with Asthma
* Being diagnosed with C.O.P.D.
* Age < 35, for the group of Young Unemployed
* Age >35 years, for the groups of Asthma and C.O.P.D. patients

Exclusion Criteria:

* Diagnosed neurological, mental or psychiatric illness
* Drug-resistance epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Neurofeedback vs. Varenicline efficacy for smoking cessation | 2 years
  The outcome measure is the effect size of each intervention measured in standardized percentage of participants that give up smoking.

SECONDARY OUTCOMES:
Effectiveness in changing quality of life as measured by EuroQL-5D | 2 years
  The outcome measure is the change from baseline in the scoring of the a questionnaire evaluating quality of life (EuroQL-5D), after the completion of the intervention.
General health | 2 years
  The outcome measure is the change from baseline in the scoring of the General Health Questionnaire which is evaluating general health, after the completion of the intervention.
Depression | 2 years
  The outcome measure is the change from baseline in the scoring of the Beck's Depression Inventory, which is evaluating depression, after the completion of the intervention.
Anxiety | 2 years
  The outcome measure is the change from baseline in the scoring of the Spielberger's State -Trait Anxiety Inventory , which is evaluating anxiety, after the completion of the intervention.
Neuroplastic effects of combined bio- and neuro- feedback training in the resting state cortical activity | 2 years
  The outcome measure is the change from baseline in the activation of the resting state cortical network after the completion of the intervention.
Neuroplastic effects of combined bio- and neuro- feedback training in the mismatch negativity response | 2 years
  The outcome measure is the change from baseline in the activation of the Mismatch Negativity response of the auditory cortex after the completion of the intervention.
Sleep quality during varenicline use | 2 years
  The outcome measure is the change from baseline in the scoring in psychometric tests evaluating sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Panos Bamidis, Ass. Prof, Principal Investigator — Medical School, Aristotle University of Thessaloniki
Locations (3):
- National Association of General Practitioners in Bulgaria, Sofia, Bulgaria
- AAI Scientific Cultural Services Ltd (AAISCS), Nicosia, Cyprus
- Laboratory of Medical Physics, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data (IPD) will be shared after obtaining the consent of the participants. The consent form will inform the participants for this attribute of the data.
  The repository will be based on popular open source software (CKAN) and it'll be accessible through a portal (endpoint) at the following address:
  ckan.smokefreebrain.eu CKAN is a powerful data management system that makes data accessible - by providing tools to streamline publishing, sharing, finding and using data. CKAN is aimed at data publishers (national and regional governments, companies and organizations) wanting to make their data open and available.
Supporting Information: Study Protocol
Time Frame: Upon completion of the study
Access Criteria: Following communication with the Principal Investigator

REFERENCES:
- [Background] Bamidis PD, Paraskevopoulos E, Konstantinidis E, Spachos D, Billis A. Multimodal e-Health Services for Smoking Cessation and Public Health: The SmokeFreeBrain Project Approach. Stud Health Technol Inform. 2017;245:5-9. PMID 29295041
- [Derived] Pandria N, Athanasiou A, Styliadis C, Terzopoulos N, Mitsopoulos K, Paraskevopoulos E, Karagianni M, Pataka A, Kourtidou-Papadeli C, Makedou K, Iliadis S, Lymperaki E, Nimatoudis I, Argyropoulou-Pataka P, Bamidis PD. Does combined training of biofeedback and neurofeedback affect smoking status, behavior, and longitudinal brain plasticity? Front Behav Neurosci. 2023 Jan 27;17:1096122. doi: 10.3389/fnbeh.2023.1096122. eCollection 2023. PMID 36778131
- See also: SmokeFreeBrain Project web-site — http://smokefreebrain.eu/
- Available data/document: Individual Participant Data Set: neurofeedback-auth — http://ckan.smokefreebrain.eu/